CLINICAL TRIAL: NCT01316965
Title: CONFUCIUS Study : Impact of a Multifaceted Program to Prevent Postoperative Delirium in the Elderly
Brief Title: Impact of a Multifaceted Program to Prevent Postoperative Delirium in the Elderly
Acronym: CONFUCIUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment of patients insufficient
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009.577
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Delirium
Keywords: Postoperative delirium; elderly; prevention; stepped wedge design; healthcare workers
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- multifaceted prevention program (Experimental)
  Interventions: Behavioral: Multifaceted prevention program HELP(Hospital Elder Life Program)
- usual care (No Intervention)

INTERVENTIONS:
Behavioral: Multifaceted prevention program HELP(Hospital Elder Life Program) — * A. Structured geriatric consultation will be performed by geriatricians of the MGT(Mobile Geriatric Teams) before surgery, including clinical examination and geriatric assessment
  * B. All members of medical and nursing staffs will attend a two hours training session performed by the MGTs and HELP(Hospital Elder Life Program) will be implemented in the surgical wards
  * C. On a quarterly basis, all members of medical and nursing staffs and MGTs will gathered to analyze medical records of patients having experienced a postoperative delirium.
  Arms: multifaceted prevention program

SUMMARY:
Postoperative delirium is common in the elderly and is associated with a significant increase in mortality, complications, length of hospital stay and admission in long care facility. Several interventions have proved their effectiveness to prevent it but their combination within a multifaceted intervention needs to be assessed using rigorous methodology based on randomized study design. CONFUCIUS trial aims to measure the impact of a multifaceted program on the prevention of postoperative delirium in elderly.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged over 75 years
* Admission for a scheduled surgery (i.e. all oncologic digestive surgery , ureterostomy, nephrectomy or cystectomy, total hip or knee replacement)
* Participation agreement

Exclusion Criteria:

* Patients with a progressive and/or poorly managed psychiatric pathology (patients with stabilized depression could be included in the study)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 175 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium rate within 7 days after surgery | 7 days after surgery

SECONDARY OUTCOMES:
Mean delirium intensity within 7 days after surgery | 7 days after surgery
Length of hospital stay | Hospital discharge
Postoperative complications 30 days after surgery incidence | 30 days after surgery
Mortality 6 months after surgery | 6 months after surgery
Feasibility of the multidisciplinary prevention program | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre KROLAK-SALMON, Pr, Principal Investigator — Hospices Civils de Lyon- Hôpital des Charpennes
Locations (1):
- Hospices Civils de Lyon-Hôpital des Charpennes, Villeurbanne, France

REFERENCES:
- [Derived] Mouchoux C, Rippert P, Duclos A, Fassier T, Bonnefoy M, Comte B, Heitz D, Colin C, Krolak-Salmon P. Impact of a multifaceted program to prevent postoperative delirium in the elderly: the CONFUCIUS stepped wedge protocol. BMC Geriatr. 2011 May 18;11:25. doi: 10.1186/1471-2318-11-25. PMID 21592324